CLINICAL TRIAL: NCT01523002
Title: Open-label, Drug Interaction Study of Pyronaridine-artesunate and Metoprolol in Healthy Volunteers and Pyronaridine-artesunate Redosing Study in Healthy Volunteers
Brief Title: Drug Interaction Study of Pyronaridine-artesunate & Metoprolol, & Redosing Study of Pyronaridine-artesunate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-014-11
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Malaria
Keywords: pyronaridine artesunate (Pyramax); artemisinin based combination therapy (ACT); metoprolol; drug-drug interaction study; redosing study
MeSH Terms: conditions — Malaria | interventions — Metoprolol; pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: metoprolol and pyronaridine-artesunate 90-day redosing (Active Comparator): Subjects will take 1 day of metoprolol followed by a 7 day wash out period, then 2 days of pyronaridine-artesunate followed by 1 day of pyronaridine-artesunate + metoprolol, followed by a 87 day follow-up period. Subjects will then receive pyronaridine-artesunate once daily for 3 days followed by a 40 day follow-up period.
  Interventions: Drug: Metoprolol and pyronaridine-artesunate
- Arm B: pyronaridine-artesunate 60-day redosing (Active Comparator): Subjects will take pyronaridine-artesunate once daily for 3 days, followed by a 57 day follow-up period. Subjects will then take pyronaridine-artesunate once daily for 3 days followed by a 40 day follow-up period.
  Interventions: Drug: pyronaridine-artesunate

INTERVENTIONS:
Drug: Metoprolol and pyronaridine-artesunate — On Day 1, subjects will receive a single oral 100 mg dose of metoprolol tartrate. On Day 8 and Day 9, subjects will receive a once daily oral dose of pyronaridine-artesunate as follows:
  55 - < 65 kg: 3 tablets (180:60 mg pyronaridine:artesunate)
  ≥ 65 kg: 4 tablets (180:60 mg pyronaridine:artesunate)
  On Day 10, a 100 mg dose of metoprolol will be coadministered with pyronaridine-artesunate at the above dose.
  On Days 98 - 100, subjects will receive pyronaridine-artesunate once daily at the same dose described above. Followed by a 40 day follow-up period.
  Arms: Arm A: metoprolol and pyronaridine-artesunate 90-day redosing
Drug: pyronaridine-artesunate — On Days 1 to 3, subjects will receive 3 days of pyronaridine-artesunate as follows:
  55 - < 65 kg: 3 tablets (180:60 mg pyronaridine:artesunate)
  ≥ 65 kg: 4 tablets (180:60 mg pyronaridine:artesunate)
  On Days 61 to 63, subjects will be redosed with a 3 day course of pyronaridine-artesunate at the above dose.
  Followed by a 40 day follow-up period.
  Other Names: Pyramax
  Arms: Arm B: pyronaridine-artesunate 60-day redosing

SUMMARY:
The primary objective of the drug-drug interaction study is to evaluate any drug interaction between the CYP2D6 substrate metoprolol and pyronaridine-artesunate in healthy volunteers.

The primary objective of the pyronaridine-artesunate redosing study is to determine the safety of redosing a 3-day regimen of pyronaridine-artesunate following 60 or 90 days in healthy volunteers.

DETAILED DESCRIPTION:
This was a phase I, open-label, randomised, 2-arm parallel group study in healthy subjects. The study population will include 44 healthy subjects (22 per treatment arm), comprising male and female adults (18-55 years) of any ethnic origin.

Subjects will be randomised to either Arm A or Arm B. Arm A will evaluate pyronaridine-artesunate interference on metoprolol pharmacokinetics (PK) and the effect of a 90-day (±7 days) redosing interval on the safety profile of pyronaridine-artesunate. Arm B will evaluate the effect of a 60-day (±7 days) redosing interval on the safety profile of pyronaridine-artesunate.

Screening will be performed in the 14-day period prior to the first dose. In Arm A, each subject will partake in 3 inpatients periods between: Days -1 to 2, Days 7 to 11, and Days 97 to 101, with dosing on Days 1, 8 to 10, and 98 to 100. In Arm B, each subject will partake in 2 inpatient periods: Days -1 to 4 and Days 60 to 64, with dosing on Days 1 to 3 and 61 to 63. Subjects will be considered to have completed the study at Day 140 (Arm A) or at Day 103 (Arm B).

Any adverse event ongoing at the time of study completion will be followed until resolution unless no further change is expected according to the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18 and 55 years with a body weight between 50 and 90 kg and a body mass index calculated using Quetelet's Index - weight (kg)/height2 (m2) between 18.5-30.0
2. Signed and dated a written informed consent form before undergoing any study related activities
3. Medically normal subjects with no significant abnormal findings at the screening physical examination as evaluated by the investigator
4. Strictly normal values of alanine aminotransferase, aspartate aminotransferase, and total bilirubin and normal or abnormal and clinically insignificant results of the other blood and urine laboratory parameters at screening.
5. Female subjects of non-childbearing potential (i.e. physiologically incapable of becoming pregnant, including any female who was post-menopausal (i.e. one year without menses) or who has undergone sterilization (via hysterectomy or bilateral tubal ligation)
6. Female subjects of childbearing potential with a negative urine pregnancy test at screening confirmed at Day -1 by a serum pregnancy test and who agreed to one of the following methods:

   * Double barrier method of contraception for 2 weeks before first study drug administration and throughout the entire study follow up period
   * Partner(s) who had undergone vasectomy and has been negative for sperm for at least 6 months
7. The ability to understand the requirements of the study and willingness to comply with all study procedures

Exclusion Criteria:

1. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, acute corrected QT interval greater or equal to 450 milliseconds), respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric or other abnormality (including head trauma)
2. Known history of hypersensitivity, allergic or adverse reactions to pyronaridine or artesunate or other artemisinins or metoprolol.
3. Other contraindications to pyronaridine use
4. Other contraindications to metoprolol use including second or third degree atrioventricular block, heart rate below 50 beats per minute, uncompensated heart failure or need for treatment with inotropic agents, clinically apparent hypotension, sinus bradycardia or sick sinus syndrome, peripheral arterial disease, pheochromocytoma, asthma, chronic obstructive pulmonary disease, depression and any other condition with in the opinion of the Investigator may be worsened by administration of metoprolol.
5. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab)
6. Seropositive HIV antibody
7. Previous participation in any clinical study with pyronaridine:artesunate (Pyramax)
8. Presence or recent history (last two years) of tobacco abuse (≥10 cigarettes/day)
9. Known or suspected alcohol abuse or illicit drug use 10 years before the study start or positive findings on urine drug screen
10. Intake of alcoholic beverages within 72 hours before study drug administration or caffeine-containing food or beverages, such as coffee, tea, chocolate, or cola, 48 hours before study drug administration
11. Gilbert's disease
12. Administration of any systemic medication or herbal product within 14 days before the first dose of study drug. If the investigator considers that the specific product would not interfere with the safety of the subject or the objectives of the study, topical treatments as well as vitamins and mineral supplements not containing other substances are allowed until 4 days before each dose. Ibuprofen at doses of at most 1200 mg per day for no more than 3 consecutive days or 6 non-consecutive days is allowed until 24h before the first dose of study drug.
13. Plasma donation 3 months before the study start
14. Blood donation of 500 mL or more 3 months before the study start
15. Participation in any clinical study in last 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Pokorny, MD, MSc, Principal Investigator — Covance Research Unit AG
Locations (1):
- Covance Clinical Research Unit AG, Allschwil, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing: Subjects will take 1 day of metoprolol followed by a 7 day wash out period; then 2 days of pyronaridine-artesunate followed by 1 day of pyronaridine-artesunate + metoprolol and then a 87 day follow-up period. Subjects will then receive pyronaridine-artesunate once daily for 3 days followed by a 40 day follow-up period.
Period: Period 1
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing | Arm B: Pyronaridine-artesunate 60-day Redosing
Started (Arm A: metaprolol (Day 1) Arm B: pyronaridine-artesunate (Days 1, 2 & 3)) | 26 | 30
Completed | 24 | 19
Not Completed | 2 | 11
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 8
Period: Period 2
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing | Arm B: Pyronaridine-artesunate 60-day Redosing
Started (Arm A: pyronaridine-artesunate (Days 8 & 9); pyronaridine-artesunate and metoprolol (Day 10) Arm B: pyronaridine-artesunate (Days 61, 62 & 63)) | 24 | 19
Completed | 18 | 13
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Adverse Event | 2 | 5
Period: Period 3
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing | Arm B: Pyronaridine-artesunate 60-day Redosing
Started (Arm A: Pyronaridine-artesunate (Days 98, 99 & 100) Arm B: NA for study design) | 18 | 0 (Arm B did not participate in Period 3)
Completed | 14 | 0
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Re-dosing: Subjects will take 1 day of metoprolol followed by a 7 day wash out period; then 2 days of pyronaridine-artesunate followed by 1 day of pyronaridine-artesunate + metoprolol and then a 87 day follow-up period. Subjects will then receive pyronaridine-artesunate once daily for three days followed by a 40 day follow-up period and a study completion evaluation.
  Metoprolol and pyronaridine-artesunate: On Day 1, subjects will receive a single oral 100 mg dose of metoprolol tartrate. On Day 8 and Day 9, subjects will receive a once daily oral dose of pyronaridine-artesunate as follows:
  55 - < 65 kg: 3 tablets (180:60 mg pyronaridine:artesunate)
  ≥ 65 kg: 4 tablets (180:60 mg pyronaridine:artesunate)
  On Day 10, a 100 mg dose of metoprolol will be coadministered with pyronaridine-artesunate at the above dose.
  On Days 98 - 100, subjects will receive pyronaridine-artesunate once daily at the same dose described above.
- Arm B: Pyronaridine-artesunate 60-day Re-dosing: Subjects will take pyronaridine-artesunate once daily for 3 days, followed by a 57 day follow-up period. Subjects will then take pyronaridine-artesunate once daily for 3 days followed by a 40 day follow-up period.
  pyronaridine:artesunate: In the first period, subjects will receive 3 days of pyronaridine-artesunate as follows: 55 - < 65 kg: 3 tablets (180:60 mg pyronaridine:artesunate)
  ≥ 65 kg: 4 tablets (180:60 mg pyronaridine:artesunate) followed by a 57 day follow-up period. In the second period, subjects will receive 3 days of pyronaridine-artesunate at the dose described above.
- Total: Total of all reporting groups
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Re-dosing | Arm B: Pyronaridine-artesunate 60-day Re-dosing | Total
Number analyzed (Participants) | 26 | 30 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (7.1) | 42 (9.4) | 43 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 13 | 16 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 24 | 30 | 54
  Black | 1 | 0 | 1
  Oriental/Asian | 1 | 0 | 1
Body weight [Mean (Standard Deviation); unit: kg] | 74.4 (11.37) | 69.8 (10.15) | 71.9 (10.88)
Height [Mean (Standard Deviation); unit: cm] | 171 (8.2) | 170 (7.4) | 171 (7.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (2.59) | 24.1 (2.67) | 24.6 (2.68)
CYP2D6 Phenotype [Count of Participants; unit: Participants]
  Poor metabolizer | 1 | 2 | 3
  Intermediate metabolizer | 11 | 13 | 24
  Extensive metabolizer | 13 | 14 | 27
  Ultra-Rapid metabolizer | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Arm A Pharmacokinetic Parameters of Metoprolol & α-hydroxymetoprolol: Area Under Curve (AUC)0-t, AUC0-∞
Description: AUC0-t & AUC0-∞ of Metoprolol & α-hydroxymetoprolol for Period 1 (metoprolol alone) & Period 2 (pyronaridine-artesunate with metoprolol)
  Abbreviations: AUC = area under the concentration-time curve; AUC0-t = AUC from Hour 0 to the last quantifiable concentration time (LQCT), where LQCT is the time at which the last sample with a quantifiable concentration was drawn; AUC0-∞ = AUC from Hour 0 to infinity
Time Frame: Plasma samples taken predose and following metoprolol dosing at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours postdose on Days 1 & 10
Population: 26 participants analyzed for Period 1, 22 participants analyzed for Period 2 (22 participants reached D10 for data collection)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/ml
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing
Number analyzed (Participants) | 26
ng.h/ml
  Period 1 AUC0-t Metoprolol | 685 (91)
  Period 1 AUC0-∞ Metoprolol | 746 (89)
  Period 2 AUC0-t Metoprolol: number analyzed (Participants) | 22
  Period 2 AUC0-t Metoprolol | 895 (77.0)
  Period 2 AUC0-∞ Metoprolol: number analyzed (Participants) | 22
  Period 2 AUC0-∞ Metoprolol | 958 (77.3)
  Period 1 AUC0-t α-hydroxymetoprolol | 707 (51.6)
  Period 1 AUC0-∞ α-hydroxymetoprolol | 804 (41.9)
  Period 2 AUC0-t α-hydroxymetoprolol: number analyzed (Participants) | 22
  Period 2 AUC0-t α-hydroxymetoprolol | 601 (72.2)
  Period 2 AUC0-∞ α-hydroxymetoprolol: number analyzed (Participants) | 22
  Period 2 AUC0-∞ α-hydroxymetoprolol | 739 (49.5)

2. Primary Outcome: Arm A Pharmacokinetics Parameters of Metoprolol & α-hydroxymetoprolol: Tmax
Description: tmax of Metoprolol & α-hydroxymetoprolol for Period 1 (metoprolol alone) & Period 2 (pyronaridine-artesunate with metoprolol)
  Abbreviations: tmax = time to maximum observed concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing
Number analyzed (Participants) | 26
hours
  Period 1 tmax Metoprolol | 1.5 [0.75 to 3.00]
  Period 2 tmax Metoprolol: number analyzed (Participants) | 22
  Period 2 tmax Metoprolol | 1.00 [0.75 to 2.02]
  Period 1 tmax α-hydroxymetoprolol | 1.5 [0.75 to 8.00]
  Period 2 tmax α-hydroxymetoprolol: number analyzed (Participants) | 22
  Period 2 tmax α-hydroxymetoprolol | 1.5 [0.42 to 6.00]

3. Primary Outcome: Arm A Pharmacokinetics Parameters of Metoprolol & α-hydroxymetoprolol: t1/2
Description: t1/2 of Metoprolol & α-hydroxymetoprolol for Period 1 (metoprolol alone) & Period 2 (pyronaridine-artesunate with metoprolol)
  Abbreviations: t1/2 = apparent terminal phase half-life
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing
Number analyzed (Participants) | 26
hours
  Period 1 t1/2 Metoprolol | 3.39 (24.78)
  Period 2 t1/2 Metoprolol: number analyzed (Participants) | 22
  Period 2 t1/2 Metoprolol | 3.28 (30.3)
  Period 1 t1/2 α-hydroxymetoprolol | 7.34 (30.8)
  Period 2 t1/2 α-hydroxymetoprolol: number analyzed (Participants) | 22
  Period 2 t1/2 α-hydroxymetoprolol | 7.55 (29.3)

4. Primary Outcome: Arm A Pharmacokinetics Parameters of Metoprolol & α-hydroxymetoprolol: Cmax
Description: Cmax of Metoprolol & α-hydroxymetoprolol for Period 1 (metoprolol alone) & Period 2 (pyronaridine-artesunate with metoprolol)
  Abbreviations: Cmax = maximum peak observed concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing
Number analyzed (Participants) | 26
hours
  Period 1 Cmax Metoprolol | 152.7 (77.1)
  Period 2 Cmax Metoprolol: number analyzed (Participants) | 22
  Period 2 Cmax Metoprolol | 228.6 (62.3)
  Period 1 Cmax α-hydroxymetoprolol | 73.9 (75.9)
  Period 2 Cmax α-hydroxymetoprolol: number analyzed (Participants) | 22
  Period 2 Cmax α-hydroxymetoprolol | 66.8 (78.4)

5. Primary Outcome: World Health Organization (WHO) Treatment Emergent Adverse Events
Description: To assess the safety of redosing a 3-day regimen of pyronaridine-artesunate. Grade 1: mild adverse event Grade 2: moderate adverse event Grade 3: severe and undesirable adverse event Grade 4: life threatening adverse event Grade 5: fatal adverse event resulting in death
Time Frame: 140 days
Measure: Number; unit: participants
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing | Arm B: Pyronaridine-artesunate 60-day Redosing
Number analyzed (Participants) | 26 | 30
participants
  Grade 1 toxicity | 25 | 24
  Grade 2 toxicity | 12 | 17
  Grade 3 toxicity | 2 | 4
  Grade 4 toxicity | 0 | 2

6. Primary Outcome: Non-WHO Listed Treatment Emergent Adverse Events
Description: To assess the safety of redosing a 3-day regimen of pyronaridine-artesunate
Time Frame: 140 days
Measure: Number; unit: participants
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing | Arm B: Pyronaridine-artesunate 60-day Redosing
Number analyzed (Participants) | 26 | 30
participants
  Mild | 23 | 21
  Moderate | 5 | 14
  Severe | 0 | 0
  Life-threatening | 0 | 0

ADVERSE EVENTS:
Time Frame: Arm A: 140 days + follow up if necessary Arm B: 103 days + follow up if necessary
Description: An adverse event is defined as any unfavourable and unintended sign, symptom, syndrome, or illness that developed or worsened during the period of observation in the clinical study.
  Clinically relevant abnormal results of diagnostic procedures including abnormal laboratory findings which are considered by the Investigator to be detrimental should be recorded as adverse events whether or not they have a causal relationship with the study drug.
Groups:
- Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing: Subjects will take 1 day of metoprolol followed by a 7 day wash out period; then 2 days of pyronaridine-artesunate followed by 1 day of pyronaridine-artesunate + metoprolol and then a 87 day follow-up period. Subjects will then receive pyronaridine-artesunate once daily for three days followed by a 40 day follow-up period and a study completion evaluation.
Arm/Group | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing | Arm B: Pyronaridine-artesunate 60-day Redosing
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/30
Other Adverse Events (participants affected / at risk) | 25/26 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing (N=26) | Arm B: Pyronaridine-artesunate 60-day Redosing (N=30)
Exanthema (rash) (Skin and subcutaneous tissue disorders) | 0 | 1 (3)
Discus hernia (intervertebral disc protrusion) (Musculoskeletal and connective tissue disorders) | 0 | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Metoprolol DDI and Pyronaridine-artesunate 90-day Redosing (N=26) | Arm B: Pyronaridine-artesunate 60-day Redosing (N=30)
Diarrhoea (Gastrointestinal disorders) | 20 (66) | 18 (58)
Nausea (Gastrointestinal disorders) | 12 (18) | 11 (13)
Vomiting (Gastrointestinal disorders) | 5 (5) | 9 (12)
Abdominal pain (Gastrointestinal disorders) | 6 (10) | 6 (10)
Abdominal pain discomfort (Gastrointestinal disorders) | 3 (5) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 2 (2)
Flatulence (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (17) | 16 (22)
Aspartate aminotransferase increased (Investigations) | 8 (9) | 17 (20)
Gamma-glutamyltransferase increased (Investigations) | 5 (7) | 14 (17)
Neutrophil count decreased (Investigations) | 2 (5) | 3 (7)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (3) | 1 (1)
Prothrombin time prolonged (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 15 (33) | 16 (24)
Dizziness (Nervous system disorders) | 9 (11) | 6 (7)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 10 (13) | 5 (6)
Chills (General disorders) | 1 (2) | 2 (2)
Malaise (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Vessel puncture site (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasopharngitis (Infections and infestations) | 3 (3) | 6 (6)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 5 (5) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No